CLINICAL TRIAL: NCT03311607
Title: Safety and Effectiveness of Short-course AmBisome in the Treatment of Post-Kala-azar Dermal Leishmaniasis (PKDL): a Prospective Cohort Study in Bangladesh
Brief Title: Safety and Effectiveness of Short-course AmBisome in the Treatment of PKDL in Bangladesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSF PKDL STUDY
Record Dates: First submitted 2017-10-03; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Post-kala-azar Dermal Leishmaniasis
Keywords: Post-kala-azar Dermal Leishmaniasis; Visceral Leishmaniasis; AmBisome; Liposomal amphotericin B; Bangladesh; Kala azar
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cohort treated with AmBisome 15 mg/kg (Other): 280 patients, receiving AmBisome
  Interventions: Drug: AmBisome

INTERVENTIONS:
Drug: AmBisome — A total dose of 15 mg/kg AmBisome given in doses of 3 mg/kg in a biweekly dosing schedule

SUMMARY:
The safety and effectiveness of AmBisome 15 mg/kg, given over 15 days in 5 biweekly infusions of 3 mg/kg on an outpatient basis, is evaluated in clinically diagnosed PKDL patients of 12 years and older in a highly endemic area in Bangladesh. This is a prospective study, with the objective to assess final cure 12 months after treatment.

DETAILED DESCRIPTION:
The safety and effectiveness of AmBisome 15 mg/kg, given over 15 days in 5 biweekly infusions of 3 mg/kg on an outpatient basis, was evaluated in clinically diagnosed PKDL patients of 12 years and older in a highly endemic area in Bangladesh. This was a prospective study, with the objective to assess final cure 12 months after treatment. Clinical response was monitored at 1, 3, 6, and 12 months after treatment, and safety during and up until one month after treatment. A total of 280 patients recruited between 8 April and 25 November 2014 received AmBisome. Of these, 272 were assessed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

-Patients of 12 years and older with probable PKDL (skin lesions strongly suggestive of PKDL with exclusion of other skin diseases, a history of VL treatment and a positive serological rK39 test)

Exclusion Criteria:

* PKDL and concurrent VL
* Prior treatment for PKDL
* On medication with a side effect profile overlapping with that of AmBisome
* A known hypersensitivity to AmBisome
* Pregnant and lactating women,
* Known cardiac disease, hepatic impairment or another severe chronic underlying disease -Renal impairment (baseline serum creatinine > 1.3 mg/dL)
* Serum potassium <3.5mmol/L at baseline

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2015-10-14 (Actual)

PRIMARY OUTCOMES:
Final outcome | 12 months
  The final outcome at 12 months was scored after carefully visual evaluation of the progress of all lesions of each patient compared to baseline.

SECONDARY OUTCOMES:
Safety | 7 weeks
  Adverse events and serious adverse events were recorded during and up to one month after treatment.
Hypokalaemia | 7 weeks
  Assessment of hypokalaemia was based on serum potassium, measured in blood samples taken at different times during and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Koert Ritmeijer, PhD, Study Director — Medecins Sans Frontieres, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided